CLINICAL TRIAL: NCT00872716
Title: Anxiolytic Effects of Single-dose Quetiapine XR Administration on Clinical Symptoms and Amygdala Activation During Exposure in Patients With Simple Phobia
Brief Title: Quetiapine in Specific Phobia
Acronym: QUISS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Prof. Dr. med. P. Zwanzger, University Hospital Muenster
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: D1443L00051; EudraCT-Nr: 2008-001371-30
Record Dates: First submitted 2009-03-30; First posted 2009-03-31 (Estimated); Last update posted 2011-03-31 (Estimated); Status verified 2011-03

CONDITIONS: Specific Phobia
Keywords: specific phobia; simple phobia; anxiety disorder
MeSH Terms: conditions — Phobia, Specific; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Quetiapine XR (Experimental): 100 mg single-dose Quetiapine XR
  Interventions: Drug: Quetiapine XR
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Quetiapine XR — 100 mg single-dose Quetiapine XR
  Other Names: - Seroquel XR; - Seroquel Prolong; - ATC-Code: N05A H04
  Arms: Quetiapine XR
Other: Placebo — Placebo
  Other Names: no other name
  Arms: Placebo

SUMMARY:
The study hypothesis is that quetiapine XR has anxiolytic properties. The study aims to investigate the putative anxiolytic properties of quetiapine XR in patients with anxiety disorders. Therefore, in a proof-of-concept design patients with simple phobia will be selected to investigate specific anxiolytic and antipanic activity during acute anxiety. Moreover, in a combined fMRI/visual stimulus presentation paradigm activity of fear-network associated brain structures such as the amygdala will be investigated under treatment with quetiapine XR or placebo. Additionally, genetic factors potentially mediating anxiolytic properties of quetiapine will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* A diagnosis of simple phobia by Diagnostic and Statistical Manual of Mental Disorders-Fourth Edition (DSM-IV)
* Females or males aged 18 to 70 years
* Females of childbearing potential must have a negative serum pregnancy test within 7 days prior or at enrolment and be willing to use an effective method of birth control for the duration of the study. Effective methods of birth control are defined as those which result in a low failure rate (i.e. pearl-index < 1%) when used consistently and correctly such as: a hormonal oral, transdermal, or injectable contraceptive agent with a double-barrier method; an implantable contraceptive device with a failure rate less than 1% for at least 3 months prior to enrolment; vasectomized partner
* Able to understand and comply with the requirements of the study

Exclusion Criteria:

* Pregnancy or lactation
* Any DSM-IV Axis I disorder not defined in the inclusion criteria
* Patients who, in the opinion of the investigator, pose an imminent risk of suicide or a danger to self or others
* Known intolerance or lack of response to quetiapine fumarate as judged by the investigator
* Use of any of the following cytochrome P450 3A4 inhibitors in the 14 days preceding enrolment including but not limited to: ketoconazole, itraconazole, fluconazole, erythromycin, clarithromycin, troleandomycin, indinavir, nelfinavir, ritonavir, fluvoxamine and saquinavir
* Use of any of the following cytochrome P450 3A4 inducers in the 14 days preceding enrolment including but not limited to: phenytoin, carbamazepine, barbiturates, rifampin, St. John's Wort, and glucocorticoids
* Administration of a depot antipsychotic injection within one dosing interval (for the depot) before randomization
* Substance or alcohol dependence at enrolment (except dependence in full remission, and except for caffeine or nicotine dependence), as defined by DSM-IV criteria
* Opiates, amphetamine, barbiturate, cocaine, cannabis, or hallucinogen abuse by DSM-IV criteria within 4 weeks prior to enrolment
* Medical conditions that would affect absorption, distribution, metabolism, or excretion of study treatment
* Unstable or inadequately treated medical illness (e.g. congestive heart failure, angina pectoris, hypertension) as judged by the investigator
* Involvement in the planning and conduct of the study
* Previous enrolment or randomization of treatment in the present study.
* Participation in another drug trial within 4 weeks prior enrolment into this study or longer in accordance with local requirements
* A patient with Diabetes Mellitus (DM) fulfilling one of the following criteria: Unstable DM defined as enrolment glycosylated hemoglobin (HbA1c) >8.5%; Admitted to hospital for treatment of DM or DM related illness in past 12 weeks; Not under physician care for DM; Physician responsible for patient's DM care has not indicated that patient's DM is controlled; Physician responsible for patient's DM care has not approved patient's participation in the study; Has not been on the same dose of oral hypoglycaemic drug(s) and/or diet for the 4 weeks prior to randomization. For thiazolidinediones (glitazones) this period should not be less than 8 Weeks; Taking insulin, if the daily dose on one occasion in the past 4 weeks has been more than 10% above or below their mean dose in the preceding 4 weeks. Note: If a diabetic patient meets one of these criteria, the patient is to be excluded even if the treating physician believes that the patient is stable and can participate in the study.
* An absolute neutrophil count (ANC) of <= 1.5 x 109 per liter
* Exclusion criteria for magnetic resonance imaging procedures: cardiac pacemaker or defibrillator; injured by a metallic object that was NOT removed; cochlear (ear) implants; surgery involving a metallic implant (e.g. knee replacement); weight more than 300 lbs/136 kg (weight limit for scanner bed); Intra-Uterine Device (IUD); claustrophobia.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-04; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
VAS-Anxiety | on study day

SECONDARY OUTCOMES:
State-Trait-Anxiety-Inventory (STAI) | on study day
Beck Anxiety Inventory (BAI) | on study day
Phobia specific questionnaire | on study day
Acute Panic Inventory (API) | on study day
Profile of Mood States (POMS) | on study day
VAS-Avoidance | on study day
VAS-Tension | on study day
VAS-Sedation | on study day
amygdala reactivity | on study day

CONTACTS AND LOCATIONS:
Overall Officials: Peter M Zwanzger, Prof Dr med, Principal Investigator — University Hospital Muenster
Locations (1):
- University Hospital Muenster, Department of Psychiatry, Münster, Germany